CLINICAL TRIAL: NCT06331871
Title: Effectiveness of Ultrasound-Guided Percutaneous Electrical Nerve Stimulation (PENS) for Patients With Post-surgical Shoulder Pain: A Randomized Clinical Trial
Brief Title: Effectiveness of Ultrasound-Guided Nerve Stimulation for Patients With Post-surgical Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Mario Jesus Abril Servan, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004202111621
Record Dates: First submitted 2024-02-24; First posted 2024-03-26 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Ultrasound-Guided Percutaneous Electrical Nerve Stimulation
Keywords: PENS; Ultrasound; Axilar nerve; Supraescapular nerve; Shoulder; Postsurgery pain

STUDY DESIGN:
Intervention Model Description: 70 patients with shoulder pain undergoing arthroscopic surgery were recruited. They were divided into two groups at random; physiotherapy protocol group (n=35) and experimental group to which the same protocol was practiced and two sessions of ultrasound-guided percutaneous nerve stimulation (US-PENS) were added (n=35).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound-guided percutaneous nerve stimulation (US-PENS) and physiotherapy protocol. (Experimental): Ultrasound Guied Percutaneus Electrical Nerve Stimulation on the suprascapular nerve and axillary nerve, along with a manual physical therapy protocol in patients with pain and lack of function after a shoulder surgery.
  Interventions: Procedure: Ultrasound Guied Percutaneus Electrical Nerve Stimulation (US-PENS) and Manual physiotherapy protocol based on available evidence.
- Physiotherapy protocol. (Active Comparator): Only a physiotherapy protocol based on available evidence, applied to patients with pain undergoing shoulder surgery.
  Interventions: Procedure: Manual physiotherapy protocol based on available evidence.

INTERVENTIONS:
Procedure: Ultrasound Guied Percutaneus Electrical Nerve Stimulation (US-PENS) and Manual physiotherapy protocol based on available evidence. — Intervention performed by needling in the vicinity of the peripheral nerves of the shoulder under ultrasound-guided control.
  Arms: Ultrasound-guided percutaneous nerve stimulation (US-PENS) and physiotherapy protocol.
Procedure: Manual physiotherapy protocol based on available evidence. — Physiotherapy treatment based on the best scientific evidence available, based on manual therapy and passive and active kinesitherapy
  Arms: Physiotherapy protocol.

SUMMARY:
The aim of this clinical trial was to demonstrate the effectiveness of the application of ultrasound-guided percutaneous nerve stimulation (US-PENS) directed at the axillary nerve and the suprascapular nerve, in patients with post-surgical shoulder pain.

This is a randomized, longitudinal, prospective and quasi-experimental clinical trial in which a total of 70 patients divided into two groups; physiotherapy protocol group (n=35) and experimental group to which the same protocol was practiced and a US-PENS session was added (n=35).

The intervention and follow-up period of the participants took place over 12 weeks.

DETAILED DESCRIPTION:
The objective of this clinical trial is to evaluate the effects of including ultrasound-guided percutaneous nerve stimulation (US-PENS) on the suprascapular nerve and axillary nerve, along with a manual physical therapy protocol in patients with pain and lack of function after a shoulder surgery.

Methods: 70 patients with shoulder pain undergoing arthroscopic surgery were recruited.

They were divided into two groups at random; physiotherapy protocol group (n=35) and experimental group to which the same protocol was practiced and two sessions of US-PENS were added (n=35).

A series of variables were evaluated:

Pain, disability and functional impotence with the help of the NSPR, SPADI and DASH scales.

In turn, goniometry, dynamometry and calculation of the pressure pain threshold were performed.

The intervention and follow-up period of the participants lasted 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery using arthroscopic techniques for rotator cuff repair, shoulder instability injuries or arthrolysis;
* Be between the 4th and 6th week after surgery;
* Presence of pain and restriction in shoulder joint mobility in at least one of the movements analyzed after surgery;
* Patients without previous surgery on the shoulder girdle.

Exclusion Criteria:

Having undergone previous physiotherapy treatment for the same reason;

* Having undergone previous physiotherapy treatment for the same reason;
* Belonephobia and/or electrophobia;
* Pharmacological treatment with antiplatelet agents;
* Patients infiltrated with corticosteroids and/or anesthetics after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
The Numeric Pain Rating Scale (NPRS) | 12 WEEKS
  The Numeric Pain Rating Scale (NPRS) is a unidimensional, outcome measure of pain intensity in adults, including those with chronic pain due to rheumatic diseases.
  The NPRS is a segmented numerical version of the visual analog scale (VAS) in which a respondent selects a whole number between zero and ten that best reflects the intensity of their pain.
  The common format is a horizontal bar or line, and like the VAS, the NPRS is based on terms that describe the extremes of pain severity.
  Therefore, the numerical rating scale consists of 11 points (NPRS), where values close to 0 reflect less pain and values close to 10 reflect greater pain.
Disabilities of the Arm, Shoulder and Hand (DASH) | 12 WEEKS
  This is a questionnaire that determines the degree of disability in the arm, shoulder and hand, providing the evaluator with a specific outcome measure of the upper extremity.
  The questionnaire consists of 30 questions that are divided into several items: 21 of them evaluate a module on physical status, 6 on painful symptoms, and 3 final questions explore the patient's social environment. The sum of the scores for each of the items is used to calculate a final value that ranges from 0 (no disability) to 100 (most severe disability).

SECONDARY OUTCOMES:
The Shoulder Pain and Disability Index (SPADI) | 12 WEEKS
  The Shoulder Pain and Disability Index (SPADI) was developed to measure shoulder pain and disability in both primary care with mixed diagnosis and surgical patient populations, including rotator cuff injuries, adhesive capsulitis, replacement surgery or shoulder prosthesis and in a large population study of painful shoulder symptoms.
  SPADI is a self-completed questionnaire with 13 items that evaluate the level of pain and the degree of difficulty with activities of daily living in the use of the upper extremities. The pain subscale is made up of 5 items and the disability subscale is made up of 8.
  The reliability of SPADI provides an average intraclass correlation coefficient of 0.89 (ICC 0.66-0.95) and a 95% CI. A Spanish version is available that demonstrated satisfactory psychometrics in populations with different shoulder disorders.
GONIOMETRY | 12 WEEKS
  Measuring the joint ranges in each plane of the joint.
DINAMOMETRY | 12 WEEKS
  assessment of muscle strength has been and is a necessity in the physiotherapy diagnosis process. Knowing this physical capacity allows us to evaluate the functional state of a muscle and, in turn, locate dysfunctions and quantify the improvement in recovery processes.
PRESSURE PAIN THRESHOLD | 12 WEEKS
  The pressure pain threshold is defined as the amount of pressure applied to a point on a subject who is first experiencing a change from the sensation of pressure to the sensation of pain.

CONTACTS AND LOCATIONS:
Overall Officials: JOSE LU ARIAS BURIA, Study Director — Fisioterapia, Terapia Ocupacional, Rehabilitación y Medicina Física/URJC/ Fac. de CC. de la Salud; CESAR FERNÁNDEZ DE LAS PEÑAS, Study Director — Fisioterapia, Terapia Ocupacional, Rehabilitación y Medicina Física/URJC/ Fac. de CC. de la Salud
Locations (1):
- Clinica Cemtro, Madrid, Madrid, Spain